CLINICAL TRIAL: NCT00001465
Title: Characterization of the Pathogenesis of Lymphangioleiomyomatosis (LAM)
Brief Title: Study of the Disease Process of Lymphangioleiomyomatosis
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950186; 95-H-0186
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-16

CONDITIONS: Lung Disease; Pneumothorax; Tuberous Sclerosis; Lymphangioleiomyomatosis
Keywords: Smooth Muscle Proliferation; Bronchoscopy; Female; Pneumothorax; Tuberous Sclerosis; Natural History
MeSH Terms: conditions — Lung Diseases; Pneumothorax; Tuberous Sclerosis; Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAM: Patients with tissue diagnosis of LAM may be admitted for evaluation every six months, or as deemed necessary for research
  Interventions: Device: Toshibia Aquilion One CT

INTERVENTIONS:
Device: Toshibia Aquilion One CT — The Toshiba Aquilion ONE CT system is currently being used for studies in both general CT radiology and CT cardiac imaging. One of the unique aspects of the Aquilion ONE CT system is its ability to acquire whole organ volume images in a single rotation by utilizing an x-ray detector that is configured as 320 detector rows with a 0.5 mm width, providing a z-axis coverage of 16 cm of anatomy. In line with the evolutionary changes to CT systems, the Aquilion ONE will be upgraded with new technology that will expand its capabilities. The changes being made to the Aquilion ONE will provide enhancements to image acquisition capabilities, reduce ionizing radiation dose, and improve subject access to the system. All of these features assist in enhancing the safety of the currently installed Aquilion ONE CT system.

SUMMARY:
Pulmonary lymphangioleiomyomatosis (LAM) is a destructive lung disease typically affecting women of childbearing age. Currently, there is no effective therapy for the disease and the prognosis is poor.

This study is designed to determine the disease processes involved at the level of cells and molecules, in order to develop more effective therapy.

Researchers intend to identify the proteins and genes that contribute to the process of lung destruction in affected individuals.

DETAILED DESCRIPTION:
Individuals with pulmonary lymphangioleiomyomatosis develop severe destructive lung disease. Most of them are females of childbearing age. Currently, there is no proven effective therapy and the prognosis is variable. This study is designed to (a) define the clinical course of the disease and (b) elucidate the pathogenesis of the disease at the cellular and molecular levels, in order to develop more effective therapy. To accomplish this, we intend to identify the proteins and genes that contribute to the process of lung destruction in affected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

General admission criteria for patients include one or both of the following:

Findings on lung biopsy diagnostic of LAM;

Findings on chest x-ray and/or chest computed axial tomography consistent with LAM.

Patients with TSC and pulmonary LAM will be included in the study.

Normal non-smokers in the control group are defined as individuals who have not smoked for greater than or equal to 1 year and have no systemic or pulmonary disease.

Normal smokers defined as individuals with no systemic or pulmonary disease, who have smoked for greater than or equal to 1 year and have normal chest x-ray and normal pulmonary function tests may be included if needed as controls for a similar population of patients with LAM.

Pregnant and or nursing women can be included in accordance with Federal Regulations at Subpart B of 45 CFR 46 Subjects who are pregnant and or nursing will be excluded from procedures during their pregnancy that are greater than minimal risk, until they are no longer pregnant and/or nursing. Procedures that will not be completed while the subject is pregnant and/or nursing including: PFTs, Six Minute Walk Test, thoracentesis, bronchoscopy, and measurements with imaging modalities requiring contrast or with radiation exposure such as Chest x-ray, CT scan, MRI, bone densitometry (DEXA). Allowing subjects to be included in the study may glean important information about individuals with uncommon pulmonary disease during and post pregnancy.

EXCLUSION CRITERIA:

Exclusion criteria for patients include:

Age less than 16.

Advanced stage of a pulmonary or a systemic illness in which the risk of the study is judged to be significant even in the absence of a clear contraindication to the procedures.

Exclusion criteria for patients for the formal exercise study and the stress echocardiogram include patients on continuous oxygen. Patients may perform an exercise test that will assess the patient's exercise capacity with activities of daily living.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with pulmonary lymphangioleiomyomatosis develop severe destructive lung disease. Most of them are females of childbearing age. This study is designed to (a) define the clinical course of the disease and (b) elucidate the pathogenesis of the disease at the cellular and molecular levels, in order to develop more effective therapy. To accomplish this, we intend to identify the proteins and genes that contribute to the process of lung destruction in affected individuals.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1995-12-18 (Actual)

PRIMARY OUTCOMES:
Define the clinical course of the disease LAM andelucidate the pathogenesis of LAM at cellular and molecular levels | on going
  To define the molecular basis of the remarkable proliferation of immature appearing smooth muscle cells, which is the cause of many of the clinical manifestations, and perhaps thereby to improve our understanding of the mechanism of smooth muscle cell proliferation in other diseases, e.g., interstitial lung diseases, asthma, atherosclerosis, hypertension, and post-angioplastic coronary restenosis. To assess the contribution of proteins and genetic factors to cyst formation, airway obstruction, and clinical course. To evaluate the role of TSC genes in the pathogenesis of LAM.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Matthew BP, Lebron A, Chen YC, Lohr WH, Rollison SF, Worthy TA, Jones AM, Julien-Williams P, Pirooznia M, Chen MY, Moss J, Wen H. Novel Pulmonary Cyst Characteristics Associated with the Diffusing Capacity of the Lung in Lymphangioleiomyomatosis: A Cross-Sectional Clinical Trial. Ann Am Thorac Soc. 2023 Jul;20(7):1073-1076. doi: 10.1513/AnnalsATS.202212-1003RL. No abstract available. PMID 36930738
- [Derived] Matthew BP, Hasani AM, Chen YC, Pirooznia M, Stylianou M, Rollison SF, Machado TR, Quade NM, Jones AM, Julien-Williams P, Taveira-DaSilva A, Chen MY, Moss J, Wen H. Ultra-Small Lung Cysts Impair Diffusion Without Obstructing Air Flow in Lymphangioleiomyomatosis. Chest. 2021 Jul;160(1):199-208. doi: 10.1016/j.chest.2021.01.077. Epub 2021 Feb 5. PMID 33549601
- [Derived] Hu-Wang E, Schuzer JL, Rollison S, Leifer ES, Steveson C, Gopalakrishnan V, Yao J, Machado T, Jones AM, Julien-Williams P, Moss J, Chen MY. Chest CT Scan at Radiation Dose of a Posteroanterior and Lateral Chest Radiograph Series: A Proof of Principle in Lymphangioleiomyomatosis. Chest. 2019 Mar;155(3):528-533. doi: 10.1016/j.chest.2018.09.007. Epub 2018 Oct 3. PMID 30291925
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1995-H-0186.html